CLINICAL TRIAL: NCT04429750
Title: Efficacy of Intact Cord Resuscitation Compared to Immediate Cord Clamping on Cardiorespiratory Adaptation at Birth in Infants With Isolated Congenital Diaphragmatic Hernia (CDH)
Brief Title: Intact Cord Resuscitation in CDH
Acronym: CHIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018_94; 2019-A01030-57 (Other: ID-RCB number, ANSM); PHRC-18-0234 (Other: PHRC number, DGOS)
Record Dates: First submitted 2020-03-18; First posted 2020-06-12 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Rare Diseases; Congenital Diaphragmatic Hernia
Keywords: Congenital diaphragmatic hernia; resuscitation; delayed cord clamping; newborn
MeSH Terms: conditions — Rare Diseases; Hernias, Diaphragmatic, Congenital | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate umbilical cord clamping (Active Comparator): This group includes newborn infants with isolated CDH who will benefit from the standardized CDH management procedure as described in the French national CDH management guidelines ("Programme National de Soins").The resuscitation maneuvers are started after the umbilical cord is clamped.
  Interventions: Procedure: Immediate umbilical cord clamping
- Intact cord resuscitation (Experimental): This group includes newborn infants with isolated CDH who will benefit from the standardized CDH resuscitation maneuvers as described in the French national CDH management guidelines ("Programme National de Soins") before the umbilical cord is clamped. The resuscitation maneuvers are started at birth while the umbilical cord still bridges mother and child.
  Interventions: Procedure: intact cord resuscitation

INTERVENTIONS:
Procedure: Immediate umbilical cord clamping — In the immediate cord clamping group, the umbilical cord will be clamped within the first 20 seconds after birth and the infant will be transferred to the resuscitation room. The newborn infant will be intubated and mechanically ventilated as quickly as possible on the resuscitation table as recommended in the French "Programme National de Soins".
  After cardiorespiratory stabilization (i.e. heart rate>120/min, increasing preductal O2 saturation or achieving acceptable preductal SpO2 targets between 80 and 95%), the infant will be transferred to the neonatal intensive care unit (NICU). Oxytocin is infused to the mother as recommended in the local protocol (usually just after birth or cord clamping).
  Arms: Immediate umbilical cord clamping
Procedure: intact cord resuscitation — The umbilical cord will be kept intact during the initial phase of the resuscitation. The infant will be placed on a specifically designed compact trolley with a warmed platform, suitable for commencing resuscitation between the mother's legs in case of vaginal birth or near the operating table beside the mother in case of cesarean section. This trolley will be fully equipped for resuscitation, including a suction device, gas flowmeter/blender, ventilatory support, and monitoring system. Its height can be adjusted in order to position the infant close to the maternal perineum. The infant will be intubated and mechanically ventilated on this trolley. The cord will be clamped once cardiorespiratory stabilization will be obtained (i.e. heart rate>120/min, increasing preductal O2 saturation or achieving acceptable preductal SpO2 targets between 80 and 95%) or in case of spontaneous placental expulsion. The infant will be then transferred to the neonatal intensive care unit (NICU).
  Arms: Intact cord resuscitation

SUMMARY:
Isolated CDH is a rare disease (1/3500) and displays a wide range of severity and outcome. Despite attempts to standardize the management of this disease at birth and during the first months of life, the mortality varies from 20 to 50% according to different hospitals in France and abroad.

Several studies already showed the benefice of late cord clamping at birth on biological and physiological adaptation of newborns to life. Previous works also suggest a possible benefit of this procedure for babies with CDH.

This multicenter randomized clinical study aims to investigate the efficacy of intact cord resuscitation compared to immediate cord clamping on cardiorespiratory adaptation at birth in full term newborn infants with isolated CDH.

ELIGIBILITY:
Inclusion Criteria:

* Antenatal diagnosis of CDH
* No severe additional malformation or chromosomal diseases
* Full term (>36 weeks gestational age)
* No inclusion in another antenatal trial
* Written informed consents from the parents

Exclusion Criteria:

* Preterm birth less than 37 weeks gestational age
* Other severe malformation(s) or chromosomal diseases
* Twin
* Parents who may have French language understanding difficulties may not participate to the study unless they receive appropriate assistance regarding the understanding of the formal consent forms needed to get included in the study. If included in the study, regarding their French understanding level, the parents may not be proposed the auto questionnaires and interviews led by the psychologist

Ages: 36 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of infants with APGAR score < 4 at 1 min or < 7 at 5 min. | during the first ten minutes after birth
APGAR score | during the first ten minutes after birth
  APGAR at 1, 5 and 10 minutes after birth will be reassessed retrospectively by a final observer. The reassessment will be carried out using a video of the first 10 minutes of life of the newborn filmed with a camera if the parents agree. This video will only record the appearance of babies' bodies and faces

SECONDARY OUTCOMES:
Frequency of postpartum hemorrhage (PPH) defined by blood loss ≥ 500 ml | during the deliverance time
Frequency of severe PPH, defined by measured blood loss ≥ 1000 ml | during the deliverance time
Blood loss volume after birth | at 15 minutes after birth, at 1hours after birth
  the collector bag will have to be left in place at least 15 minutes to have one measure of blood loss at the same time point in all women
Frequency of infants with the need for chest compressions | during the deliverance time
Frequency of infants with the need for epinephrine administration and/or fluid resuscitation | during the deliverance time
Heart rate | at 1, 5, and 10 min after birth and at 24 hours, 48 hours, 72 hours, at 7 days and at 28 days
  a pulse oximeter sensor will be placed at the right hand as soon as possible (within the first minute after birth), which then will be connected to a pulse oximeter;
plasma lactate concentration | at one hour after birth (H1): at 24 hours, 48 hours, 72 hours, at 7 days and at 28 days
  these quantitative variables can be considered as objective markers of early cardiorespiratory adaptation at birth.
changes of global Blood gases parameters | at 1hour , 24 hours, 48 hours, 72 hours, at 7 days and at 28 days
  pre- and postductal SpO2,
changes of ventilatory parameters | at 1hour , 24 hours, 48 hours, 72 hours, at 7 days and at 28 days
  peak inspiratory pressure
changes of ventilatory parameters | at 1hour , 24 hours, 48 hours, 72 hours, at 7 days and at 28 days
  respiratory rate
Volume of fluid resuscitation | during the first 24 hours
Frequency of infants with the need for vasoactive drugs ; | during the first 24 hours
Frequency of infants with the need for pulmonary vasodilator | during the first 24 hours
Hemoglobin concentration | at 24 hours
Infant mortality rate | at 90-day after birth
Infant morbidity outcomes assessed within the first 90 days after birth | at 90-day after birth
Number of refusal of participating to the protocol. | at the end of the study period (90±7 days after birth)
  the reasons for refusal will be recorded : do not want to participate to a research protocol, to not want to be randomized in the immediate cord clamping group, to not want to be randomized in the intact cord resuscitation group;
State Trait Anxiety Inventory (STAI) revised version, form Y | within the first 48 hours after birth, and at the end of the study period (90±7 days after birth).
  The STAI is a self-report scale translated in French (1). The scale includes 20 questions, and takes approximately 5 minutes to complete. It is widely used and usually well accepted. Both parents will be requested to answer the questionnaire at two distinct moments. The first will be within the first 48 hours after birth, and the second will be during the medical consultation at the end of the study period (90±7 days after birth).
the Impact of Event Scale-Revised (IES-R) | during the 7 days prior to completion and at the end of the study period (90±7 days after birth).
  The IES-R is made up of 22 items aimed at assessing three main factors of traumatic symptoms (intrusion, avoidance and numbing, and hyperarousal) linked to a specific stressful event. The questions pertain to symptoms occurring during the 7 days prior to completion. The scale usually takes approximately 5 minutes to complete. Parents will be requested to answer the questionnaire during the medical consultation at the end of the study period (90±7 days after birth).
the Intolerance for Uncertainty Scale (EII). | at the end of the study period (90±7 days after birth).
  This self-report scale was originally designed in French and includes 27 questions pertaining to the beliefs and representations held by individuals with regards to uncertainty. The scale is usually completed in approximately 10 minutes. Parents will be requested to answer the questionnaire during the medical consultation at the end of the study period (90±7 days after birth).
Semi-structured interviews | at the end of the study period (12 months after birth)
  Semi-structured interviews will be proposed by a psychologist to the parents whatever the issue, to assess their personal experience of the resuscitating period at birth, including both early/delayed cord clamping and close/remote resuscitation maneuvers. The interviews tape recordings will be transcribed and then analyzed using thematic coding. The anonymized data will be independently coded by three researchers and compared for consistency of interpretation. The themes that emerged following the final coding will be used for a qualitative analysis of the parental verbatim; Due to he's or her's initial condition (HCD), if the newborn dies before the end of the study, the parents will not be asked to get through the psychological questionnaires and interviews
the 'faceless' acute neonatal pain scale (FANS) | during intubation
  FANS, which doesn't include items on facial expression, is particularly adapted for evaluating acute pain in newborns during intubation. Pain assessment is based on the analysis of limb movement, vocal expression and autonomic reactions, including heart rate variations and the occurrence of bradycardia or desaturation.
Cerebral Near-infrared spectroscopy recorded | at H1, H2, H6, H12, H24, H48
Echographic parameters with the Resistive index and pulsatility index in the anterior cerebral artery | at H6, H24, H24 after the chirurgical CDH repair gesture, H48, D7, D28
A parental questionnaire to assess neurological development (ASQ 3 score). | at M6 and M12

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Storme, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (3):
- France (3):
  - Chu Amiens Picardie, Amiens
  - Hop Jeanne de Flandre Chu Lille, Lille
  - Chu de Nantes -, Nantes